CLINICAL TRIAL: NCT06969638
Title: A Randomized Trial to Examine the Influence of "Likes" in Social Media Food Ads on Black and White Adolescents' Food Purchases - Study 2
Brief Title: Influence of "Likes" in Social Media Food Ads on Black and White Adolescents' Food Purchases - Study 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 20-01796-2; R01CA248441 (NIH)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: The intervention is exposure to social media food ads that are either race congruent or race incongruent, and that have varying numbers of likes.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Black Many Likes (Experimental): Food ads with many "likes" and featuring Black individuals
  Interventions: Behavioral: Black Ads; Behavioral: Many Likes
- Black Few Likes (Experimental): Food ads with few "likes" and featuring Black individuals
  Interventions: Behavioral: Black Ads; Behavioral: Few Likes
- White Many Likes (Experimental): Food ads with many "likes" and featuring White individuals
  Interventions: Behavioral: White Ads; Behavioral: Many Likes
- White Few Likes (Experimental): Food ads with many "likes" and featuring White individuals
  Interventions: Behavioral: White Ads; Behavioral: Few Likes

INTERVENTIONS:
Behavioral: Black Ads — Food ads that feature Black individuals
  Arms: Black Few Likes; Black Many Likes
Behavioral: White Ads — Food ads that feature White individuals.
  Arms: White Few Likes; White Many Likes
Behavioral: Many Likes — Food ads that have many "likes"
  Arms: Black Many Likes; White Many Likes
Behavioral: Few Likes — Food ads that have few "likes"
  Arms: Black Few Likes; White Few Likes

SUMMARY:
This is a randomized trial to examine the influence of number of "likes"on social media food ads on Black and White adolescents' food purchases

DETAILED DESCRIPTION:
The aim of this randomized trial is to test the degree to which visual attention to racially congruent vs incongruent people, and/or number of "likes" in social media ads influence Black and White adolescents' food purchases.

ELIGIBILITY:
Inclusion Criteria:

* adolescent (13-17 years of age) who identifies as only non-Latino White or only Black/African American; who logs into Instagram once daily; who can read and speak English

Exclusion Criteria:

- participants who do not meet all criteria described above.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1300 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of Calories Purchased | Day 0 (approximately 5 minutes)
  Total number of calories selected in the hypothetical snack choice pairings.

SECONDARY OUTCOMES:
Attitudes towards Ads | Day 0 (approximately 5 minutes)
  Attitudes are reported on a Likert scale of 1 to 100; higher scores indicate more positive attitudes toward the advertisements.
Engagement with Ads | Day 0 (approximately 5 minutes)
  Participants indicate in which ways, if any, they would engage with each ad by answering the following question: "How you would respond if you saw this ad on social media"? [Select all that apply: "Like" [heart icon and other emojis], comment, tag a friend, direct message a friend, re-post, none of the above]). The outcome is measured as the number of participants who indicate they would engage with ads.

CONTACTS AND LOCATIONS:
Overall Officials: Marie A. Bragg, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided